CLINICAL TRIAL: NCT06112860
Title: Over-the-counter Hearing Aids and Mild Cognitive Impairment
Brief Title: OTC Hearing Aid and MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Pamela Souza, Professor, Otolaryngology; Communication Sciences and Disorders, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU00219514
Record Dates: First submitted 2023-10-25; First posted 2023-11-02 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss; Mild Cognitive Impairment; Alzheimer Disease and Related Dementias (ADRD)
Keywords: Over-the-counter Hearing Aids
MeSH Terms: conditions — Hearing Loss; Cognitive Dysfunction; Alzheimer Disease | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Those listening and scoring recorded tasks will be blinded to which group the participants are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OTC Hearing Aid First (Other): Participants will be provided a pair of OTC hearing aids (experimental) with typical directions and use for 4 weeks before outcome measures will be assessed. After which, participants will then receive the communication strategies information/counseling (control) and have outcome measures assessed after 4 weeks.
  Interventions: Device: Over the counter hearing aid; Behavioral: Communication Strategies Information/Counseling
- Communication Strategies First (Other): Participants will receive the communication strategies information/counseling intervention (control) first. Outcome measures will be assessed at 4 weeks. After which, participants will then be given a pair of OTC hearing aids (experimental) with typical directions and use for four weeks before having outcome measures assessed.
  Interventions: Device: Over the counter hearing aid; Behavioral: Communication Strategies Information/Counseling

INTERVENTIONS:
Device: Over the counter hearing aid — An over the counter hearing aid is a device that provides amplification appropriate for individuals with mild to moderate hearing loss. Participants will receive the devices with typical directions and have one scheduled remote visit one week after receiving devices with an audiologist.
  Other Names: OTC hearing aid
Behavioral: Communication Strategies Information/Counseling — Communication Strategies provide information meant to help an individual compensate for hearing loss. The information provides tips both for the individual with hearing loss and for those communicating. People who choose not to pursue hearing aids will typically be given communication strategies information to help them manage their hearing loss. Participants will receive the counseling information in the mail and then have a 1 week follow-up appointment with an audiologist.
  Other Names: Communication Strategies

SUMMARY:
The goal of this study is to better understand if, in patients with mild to moderate hearing loss who are also experiencing mild cognitive impairment (MCI) or Alzheimer's disease and related dementias (ADRD), Over-the-Counter (OTC) hearing aids:

1. improve communication
2. Whether the magnitude of benefit depends on the patient's level of cognitive disability,
3. Whether alternative remediation (such as targeted communication strategies) offer similar benefits.

Participants and a communication partner will be randomized into an OTC first or Communication Strategies first arm, where participants will receive communication strategy information customized for those with cognitive impairment.

DETAILED DESCRIPTION:
This is a single blind cross-over study comparing OTC Hearing Aids to communication strategies information/counseling and their impact on communication between a person who has hearing loss and MCI and a communication partner. Due to the nature of the study, it will not be possible to blind the participants to which arm they are in, but the scorers will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Over 60 years of age
* Mild dementia or mild cognitive impairment. Diagnosis will be made at participating memory evaluation centers (see recruitment).
* Mild to moderate bilateral hearing loss and no current hearing aid use.
* A communication partner who is able and willing to participate in the study.
* No vision impairment that would interfere with the ability to complete study tasks (i.e., legally blind, severe cataracts, or macular degeneration)
* Able to provide own consent as evaluated by the Consent Assessment

Exclusion Criteria:

1. Clinically significant unstable or progressive medical conditions, or conditions which, in the opinion of the investigator(s) places the participant at unacceptable risk if he or she were to participate in the study.
2. History of unresolved communication difficulties following another neurological problem (i.e., stroke or brain tumor), neurodevelopmental disorder (i.e., Down's syndrome), or head/neck cancer
3. Positive history of major psychiatric disorder (i.e., schizophrenia, significant untreated depression)
4. Co-enrolled in other intervention studies targeting hearing, language, or communication strategies.
5. History or current fluctuating hearing loss

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Perception of Conversation Index - Dementia Alzheimer's Type (PCI-DAT) | Baseline at enrollment, then after 4 weeks of using each intervention
  A questionnaire completed by the communication partner of the individual with MCI and hearing loss. On this scale, higher scores reflect more frequent and more problematic conversation difficulties; item possible scores range from 0 (not problematic) to 7 (.very problematic)

SECONDARY OUTCOMES:
Hearing Handicap Inventory for the Elderly (HHIE) | Baseline at enrollment, then after 4 weeks of using each intervention
  Questionnaire has 25 items with subscales for social and emotional impacts and is scored from 0-100, with 100 representing least handicap.

OTHER OUTCOMES:
Conversation Analysis | 4 weeks after first intervention
  The Diapix conversation task where participant and communication partner find the differences in two very similar pictures by discussing them.
Adherence | 4 weeks after each intervention
  Reported Use (hours per day)
Usability | 4 weeks after OTC intervention
  We will use a modification of the Systematic Usability Scale to query the patient's experience with the OTC aids.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Souza, PhD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University HA Lab, Evanston, Illinois
  - La Crosse Mayo Clinic, La Crosse, Wisconsin
  - UW Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No